CLINICAL TRIAL: NCT00833612
Title: A Multi-center, Randomized, Controlled Study of Mechanical Left Ventricular Unloading With Counterpulsation to Reduce Infarct Size Pre-PCI for Acute Myocardial Infarction - CRISP AMI
Brief Title: Counterpulsation Reduces Infarct Size Pre-PCI for AMI
Acronym: CRISP-AMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Datascope Corp. (Industry)
Collaborators: Duke University (Other); Flinders Medical Centre (Other Government)
Responsible Party: Debra Joseph/VP Marketing and Clinical Services, Datascope Corp.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00001
Record Dates: First submitted 2009-01-27; First posted 2009-02-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: IABC; AMI
MeSH Terms: interventions — Counterpulsation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control arm of study (No Intervention)
  Interventions: Device: Counterpulsation with IAB

INTERVENTIONS:
Device: Counterpulsation with IAB — IABC pre-reperfusion PCI
  Other Names: CS100 & CS300 IAB Linear 7.5F Fidelity 8.0 F Sensation 7.0 F

SUMMARY:
Subjects with anterior acute STEMI who receive an IABC before primary PCI will have decreased MI size.

DETAILED DESCRIPTION:
Post clearance device study in which subjects with acute MI will be randomized 1:1 to either receive IAB or to receive standard of care without IAB before mechanical reperfusion. Subjects will be followed throughout their hospital stay and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an ICF
* ≥ 18 and ≤ 90 years of age
* General good health, in the opinion of the investigator
* ST elevation of 2mm in 2 contiguous anterior leads or ≥ 4mm total in anterior leads
* Scheduled for PCI < 6 hours from onset of symptoms of MI

Exclusion Criteria:

* Known contraindication to MRI
* Prior thrombolytic therapy during the index event
* Known history of MI
* Known severe aortic insufficiency
* Known aortic aneurysm
* Known severe calcific aorta-iliac disease or peripheral vascular disease
* Experiencing cardiac shock
* Known end-stage renal disease
* Weight >400 lbs. or height <4 ft.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine whether IABC before mechanical reperfusion decreases myocardial infarct (MI) size. | 3-5 days

SECONDARY OUTCOMES:
To determine the effect of IABC before mechanical reperfusion on post PCI cardiovascular function and major adverse cardiac events (MACE) (ie, death, reinfarction, and CHF) at 30 days and 6 months. | 30 days and 6 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ohman, MD, Principal Investigator — Duke University
Locations (40):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Essentia Institute of Rural Health (St Mary's), Duluth, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Newark Beth Israel Hospital, Newark, New Jersey
  - University of Rochester Medical Center-Strong Memorial Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
- Flinders Medical Centre, Bedford Park, Australia
- Virga Jesse, Hasselt, Belgium
- Institut Hospitalier Jacques Cartier, Massy, Alsace, France
- Germany (3):
  - Klinik fur Innere Medizin und Kardiologie, Dresden
  - University of Freiburg, Freiburg im Breisgau
  - Herzzentrum Leipzig GmbH, Leipzig
- India (11):
  - Gurunanak CARE Hospital, Hyderabad, Andhra Pradesh
  - Baroda Heart Institute and Research Centre, Vadodara, Gujarat
  - Saint John's Medical College and Hospital, Bangalore, Karnataka
  - Bhagwan Mahaveer Jain Heart Centre, Bangalore
  - Apollo Hospitals, Bangalore
  - Medanta - The Medicity, Delhi
  - CARE Hospital, Hyderabad
  - Tagore Hospital and Heart Care Centre, Jalandhar
  - Indraprastha Apollo Hospital, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Apollo Gleneagles Hospital, West Bengal
- Mater Misericordiae University Hospital, Dublin, Ireland
- Azienda Ospedaliero Universitaria Cargeei, Florence, Italy
- Catharina Hospital, Eindhoven, Netherlands
- United Kingdom (4):
  - Royal Bournemouth Hospital, Dorset
  - Royal Infirmary of Edinburgh, Edinburgh
  - Leeds General Infirmary, Leeds
  - St. Thomas Hospital, London

REFERENCES:
- [Derived] Patel MR, Smalling RW, Thiele H, Barnhart HX, Zhou Y, Chandra P, Chew D, Cohen M, French J, Perera D, Ohman EM. Intra-aortic balloon counterpulsation and infarct size in patients with acute anterior myocardial infarction without shock: the CRISP AMI randomized trial. JAMA. 2011 Sep 28;306(12):1329-37. doi: 10.1001/jama.2011.1280. Epub 2011 Aug 29. PMID 21878431
- [Derived] Patel MR, Thiele H, Smalling RW, Chandra P, Zhou Y, Cohen M, Perera D, Ohman EM. A multicenter, randomized, controlled study of mechanical left ventricular unloading with counterpulsation to reduce infarct size prepercutaneous coronary intervention for acute myocardial infarction: rationale and design of the Counterpulsation Reduces Infarct Size Acute Myocardial Infarction trial. Am Heart J. 2011 Jul;162(1):47-55.e1. doi: 10.1016/j.ahj.2011.03.037. PMID 21742089